CLINICAL TRIAL: NCT03022786
Title: Improving Value of Care for Patients With Severe Stasis Dermatitis
Acronym: Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Pfizer (Industry); Ohio Dermatological Association (Unknown)
Responsible Party: Principal Investigator, Susan Nedorost, Professor of Dermatology, Case Western Reserve University, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-15-10
Record Dates: First submitted 2016-12-29; First posted 2017-01-16 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Stasis Dermatitis
Keywords: Dermatitis
MeSH Terms: conditions — Dermatitis | interventions — Home Health Aides; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Understanding patient perspective (No Intervention): Patients will be interviewed who have been diagnosed with stasis dermatitis. The Principal Investigator will learn their perspective on their leg swelling, impact on quality of life, and obstacles to wearing compression stockings
- Refining tool kit (No Intervention): Using in-depth interviews for our inpatients selected using the same criteria as in Phase 1 and independent focus groups of providers, The study staff will obtain feedback to refine the items in our toolkit before implementing them in January 2017.
  There will be a focus group comprised of providers. This focus group will explore the perceptions of the providers and what unmet needs remain for the patients.
- Implementation (Other): Our patient education materials and toolkit include an order set to help providers guide patients to adhere to compression, the gold standard of care for this condition. This will also direct patients to know who to contact if itching or pain persists, what the patient can do at home, when to go to the hospital, as well as information on financial and home care assistance as it relates to managing their chronic condition.
  Interventions: Other: Order set; Other: Motivational Interviewing training for home health aides; Other: Tools & Education

INTERVENTIONS:
Other: Order set — Inpatient order set and ambulatory care guide offer guidance on initial compression to decrease edema, obtaining gradient compression stockings, how to access evaluation by vascular medicine for pain or dermatology for evaluation of allergic contact dermatitis if itch persists, etc
  Arms: Implementation
Other: Motivational Interviewing training for home health aides — Home Care aides trained about use of compression stockings and use of motivational interviewing as a tool to help patients make behavior changes to reduce leg swelling. This is part of our 'tool kit'.
  There will be a focus group comprised of providers. This focus group will explore the perceptions of the providers and what unmet needs remain for the patients.
  Arms: Implementation
Other: Tools & Education — Engaged physical therapists to evaluate patients for ability to don stockings, to assess need for strengthening exercises or leg exercises to improve venous return. This is part of our 'tool kit'
  Arms: Implementation

SUMMARY:
Explore the unmet needs of patients admitted to the hospital for severely inflamed skin of the lower legs, often described as 'bilateral cellulitis". These patients usually have intractable lower extremity edema, stasis dermatitis and sometimes allergic contact dermatitis rather than an infectious process; readmission is common. Investigators will create patient and provider education materials to align dermatological, home health, and other resources and measure reduction in hospital re-admission rate and length of stay.

DETAILED DESCRIPTION:
SPECIFIC AIMS 2.1.1 Understand the unmet needs for stasis dermatitis care from the patient and provider perspective.

PHASE 1: Patients Access problem: Severe stasis dermatitis is a multifactorial condition that can mimic "bilateral cellulitis". However, true bilateral cellulitis is exceedingly rare and in most cases, is a misdiagnosis. The diagnosis of cellulitis is based primarily on clinical appearance, sharing many features with severe stasis dermatitis. Objective measures for the diagnosis of cellulitis are rarely helpful, with low sensitivity and specificity rates for fever, leukocytosis, tachycardia, blood cultures, and imaging studies. Admissions for cellulitis and "bilateral cellulitis" in the United States are frequent, representing nearly 4% of all emergency admissions in 2010, with hospital stays averaging 5-7 days. Among the factors most highly associated with increased length of hospital stay in these patients, the top four include chronic edema, use of diuretics, elderly age, and living alone2. These patients are likely to have severe lower extremity swelling, complicating stasis dermatitis, and the most difficulty managing chronic health conditions. In a recent study of 145 patients admitted for cellulitis, it was found that 28% were incorrectly diagnosed with lower limb cellulitis, with venous stasis dermatitis being the most common diagnosis mistaken for cellulitis in 37% of cases. This is costly to patients, providers, hospitals, and the healthcare system.

In outpatient and inpatient settings, internists frequently prescribe diuretics to reduce lower extremity edema without awarding the problem a comprehensive evaluation for underlying causes. This chronic condition requires ongoing treatment, in many forms, which must address the primary cause. Gradient compression is the most effective means to achieve relief, but long-term management with this form of treatment requires a breadth of knowledge on behalf of providers and patients. For providers for example, multi-layer bandages must be used during the acute phase to reshape and reduce the size of the limb, appropriate stocking compression grade and length must be chosen, and patients and potential caregivers should be educated on donning and doffing stockings, application aids, appropriate hosiery care, skin care, use of emollients, limb massage, and exercise. Additionally, this requires stockings not covered by many insurance plans. Many patients are non-adherent because the patients do not have a family member or home health aide to assist, or the patients do not understand the importance of stockings as a treatment for the patients disease. Providers may not have knowledge of who to contact to get patients assistance in these situations. As a result, the edema gets worse, and patients are admitted and readmitted to the hospital with relapsing "bilateral cellulitis" of the lower extremities.

Phase 1 of this study was approved by the University Hospitals Institutional Review Board in January 2016 and under this protocol investigators have interviewed 27 inpatients (28 admissions) using a structured survey. The results of these interviews informed the development of a tool kit to improve care for these patients.

The tool kits consists of a patient brochure, a list of stockings and services available at local medical supply houses, and an order set that includes patient education including an Expectation Management and Medical Information (EMMI) module on compression stockings, a video patient story, and training of University Hospitals Home care aides in motivational interviewing to support adherence to regular use of gradient compression.

PHASE 2: Focus Groups Using in-depth interviews for our inpatients selected using the same criteria as in Phase 1 and independent focus groups of providers, the Principal Investigator will obtain feedback to refine the items in our toolkit before implementing them in January 2017. The focus groups will be conducted with assistance from the Clinical and Translational Science Collaborative (CTSC) Behavioral Measurement and Resource Center. The in-depth interviews will be conducted either at patient homes or as inpatients. The interviews may be recorded as in Part 1. The recordings and data will be downloaded into REDCap.

There will be a focus group comprised of providers. This focus group will explore the perceptions of the providers and what unmet needs remain for the patients. With this information, investigators will design educational materials to help align resources in a timely fashion and avoid admission when possible. The order set will include guidance on when to obtain consultations as well as specific orders for reduction of lower extremity edema and monitoring for side effects of compression.

2.1.2 Design education for patients and providers to cue them when additional care is needed.

PHASE 3: Tools & Education Access problem : Patients are often admitted to the hospital for "bilateral cellulitis" despite the fact that most of these patients do not have true skin infections. A research study published in 2015 demonstrated that 75% of inpatient dermatology consultations for 'cellulitis" resulted in a diagnosis of "pseudocellulitis" . Our data from phase 1 confirms that 75% of patients admitted for lower extremity cellulitis at University Hospitals do not in fact have cellulitis, although 90% receive antibiotics during a mean length of stay of 8.3 days. Patients and providers may not even be aware of this misdiagnosis, as stasis dermatitis will improve with leg elevation alone during a hospital stay. As a result, care givers erroneously give intravenous antibiotics all of the credit for the condition's resolution. When it recurs, a history of "recurrent cellulitis" is added to the patient's chart, and the cycle is repeated.

Providers may also struggle with a lack of objective measures that can be used in the diagnosis of cellulitis and its severity, depending primarily on clinical appearance.

Unnecessary admission and testing is expensive in many ways. For patients admitted to the hospital, standard treatment for cellulitis is IV antibiotics for a week or more. Prolonged bed rest in the hospital with potent antibiotics is problematic, especially for older patients. It puts them at risk for impaired mobility, deep venous thrombosis, nosocomial infections, particularly with Clostridium difficile, and is monetarily costly for all parties involved. Alternative diagnoses need to be considered. Allergic contact dermatitis, which is known to complicate stasis dermatitis, is one possibility. Patients can easily develop contact allergies to components of topical steroids and topical antibiotics prescribed in an attempt to treat dry, cracked, or fissured skin on an outpatient basis. However, many inpatient facilities do not have access to regular dermatological consultation, and local dermatologists may not have the appropriate patch tests or experience with patch testing to identify contact allergen in the setting of stasis dermatitis.

Patient education materials and toolkit will help patients know who to contact when the edema progresses, what patients can do at home, when to go to the hospital, as well as information on financial and home care assistance as it relates to managing chronic condition. Provider education materials will assist providers with making the correct diagnosis, ordering appropriate testing, understanding when to consider admission, especially in cases of "bilateral cellulitis", involving specialty providers, and aligning assistance for patients. The goal is to help providers when the patients feel stuck in attempting to help patients manage this chronic condition, especially after the patient has already had multiple admissions.

Measure the value of services identified in steps 1 and 2.

Investigators will track the number of patient admissions for antibiotics for "bilateral cellulitis" and length of stay at two different time points: (1) before and (2) after provider education ( e.g. clinical decision support in the electronic health record, an contact information guides for trained home health aides). Investigators will also track the number of readmissions and length of stay for patients at two time points: (1) before and (2) after patient education materials are implemented (e.g. educational brochure, information guides for community medical supply houses, and improved access e.g to increase use of patch testing for inpatients). Investigators will stratify patients who have been seen in wound care centers and those who have had patch testing and compare them to patients who have not, to help better understand the value of these services.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Inpatient admission to the hospital for inflamed skin of the lower legs, bilateral cellulitis, and contact dermatitis
* Fluent in English

Exclusion Criteria:

* Patients under the age of 18
* Illiterate patients
* Non-English speaking patients
* Outpatients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01; Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Length of stay for patients with stasis dermatitis | Up to 2 years
  Feb-Sept in both years

SECONDARY OUTCOMES:
Readmission rate for patients with stasis dermatitis | Up to 2 years
  Feb through Sept both years
Patch testing for stasis dermatitis | Up to 2 years
  Absolute number of patients referred for evaluation of secondary allergic contact dermatitis in the setting of stasis dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Susan Nedorost, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No